CLINICAL TRIAL: NCT07044518
Title: A Comparison Study: Hearing Evaluation and Real-Ear Measurements of Apple AirPods Pro 2 vs. Phonak Hearing Aids
Brief Title: The Clinical Application of Apple AirPods Pro 2 vs. Hearing Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 00005980
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hearing Loss
Keywords: hearing loss; over-the-counter hearing aid; hearing aid; OTC hearing aid
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AirPod Pro2 (Experimental)
  Interventions: Device: Over-the-Counter Hearing Aid; Device: Hearing aid, air conduction
- Hearing Aid (Active Comparator)
  Interventions: Device: Over-the-Counter Hearing Aid; Device: Hearing aid, air conduction

INTERVENTIONS:
Device: Over-the-Counter Hearing Aid — This intervention involves a self-fit, over-the-counter (OTC) hearing aid that is set up by the user with limited to no help from a hearing professional. Amplification is personalized through an app-based hearing test on a smartphone. The device is used during a single study visit (90 minutes) to assess hearing and provide amplification.
Device: Hearing aid, air conduction — This intervention uses a prescription hearing aid that is programmed and fitted based on results from a standard hearing test. The device is also used during a single study visit (90 min) for comparison purposes.

SUMMARY:
The goal of this clinical trial is to learn whether the Apple AirPods Pro 2 can accurately test hearing and provide helpful amplification, like a traditional hearing aid, in adults with hearing loss. The main questions it aims to answer are:

* Can the AirPods Pro 2 hearing test give similar results to a standard hearing test done in a sound booth by an audiologist?
* Can the AirPods Pro 2 provide amplification (make sounds louder) in a way that matches what a traditional hearing aid would provide?

Researchers will compare the AirPods Pro 2 results to standard hearing tests and hearing aid fittings to see if they perform in a similar way.

Participants will:

* Take a standard hearing test in a sound booth
* Use the Apple Hearing Test with AirPods Pro 2
* Have the loudness of the AirPods and a traditional hearing aid measured and compared using special equipment

DETAILED DESCRIPTION:
Hearing loss is becoming one of the most prevalent, yet undertreated health conditions in the United States. A staggering 5% of the world's population - or 430 million people - require rehabilitation to address their disabling hearing loss (including 34 million children), and it is estimated that by 2050, 700 million people - or 1 in every 10 people - will have disabling hearing loss (WHO, 2024). In the United States alone, the National Institute on Deafness and Other Communication Disorders predicts that approximately 15%, or 37.5 million, of American adults ages 18 years and over have some degree of hearing loss. The severity of hearing loss increases with age, affecting about one in three people between the ages of 65 and 74 years, and nearly half of those older than 75 years (NIDCD, 2023). Although hearing loss is a major health issue, it is estimated that the utilization rate of hearing aids is about 15% (Nassiri et al., 2021).

A major factor for this low utilization rate of hearing aids is the difficulty in accessibility of services for certain individuals, primarily those with financial constraints or those who live in rural areas with fewer audiologists (Carr & Kihm, 2022). Furthermore, insurance typically provides little to no coverage for hearing aids despite it being the most efficacious treatment. According to Arnold et al. (2017), Medicaid only provides hearing aid coverage in 28 states with substantial coverage variability between individual states. One way this issue has been addressed is through the development of over-the-counter hearing aids (OTCs), which can be purchased online or at a retail center without a requirement for an audiologist. The U.S. Food and Drug Administration approved the use of OTCs in 2022 for consumers 18 years or older with a perceived mild to moderate hearing loss (Stephenson, 2022). A retrospective survey study by Manchaiah et al. (2023) found that 84% of respondents expressed discomfort with OTCs and that the majority of respondents had concerns for safety, counseling, and audiological care. Although there has been some hesitation toward the use of OTCs from practicing audiologists, a study performed by Swanepoel et al. (2023) suggests that there is no significant difference in mostly objective, but also subjective, outcomes when comparing traditional hearing aids provided by hearing healthcare professionals and over-the-counter options.

A multinational tech corporation, Apple, has developed a Hearing Test Feature (HTF), an over-the-counter air-conduction hearing assessment for use with the Apple AirPods Pro 2 devices using a compatible iPhone or iPad (iOS 18.1 or higher). With their update for the AirPods Pro 2 (AP2), an individual can self-administer a hearing evaluation. The device would then use their test results, or audiogram, to set the gain in the individual's AirPods for daily use as an OTC hearing aid, using the Hearing Aid Feature (HAF). This new feature has the potential to allow users to access hearing amplification without purchasing higher-cost devices or seeing an audiologist.

Currently there is a critical gap in research that evaluates Apple's new Hearing Health Features. This project aims to research the validity of Apple's HTF and HAF by comparing results to a conventional audiologic evaluation and Phonak hearing aids.

ELIGIBILITY:
Inclusion Criteria:

* English speaking,
* Normal otoscopy
* Mild to moderate hearing loss

Exclusion Criteria:

* Non-English speaking,
* Active ear infection at time of appointment,
* Outside the normal range (score <71) on the XpressO Montreal Cognitive Assessment (MoCA)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-09-11 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Hearing evaluation | From the beginning to the end of a single study visit lasting approximately 45 minutes
  measure that evaluates hearing threshold at octave frequencies between 250 to 8000Hz; measured in dB HL.
Real Ear Measures | From the beginning to the end of a single study visit lasting approximately 45 minutes
  measures how much sound level (gain) a hearing aid is delivering at octave frequencies between 250 to 8000 Hz; measured in dB SPL.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Arizona Hearing Clinic, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No